CLINICAL TRIAL: NCT05329857
Title: Randomized, Open Label, Two-sequence, Two-treatment, Two-period, Crossover, Single Dose Bioequivalence Study Fixed-dose Combination of Metformin and Vildagliptin Tablets 1000/50 mg Manufactured by Oman Pharmaceuticals Products Co. LLC, Sultanate of Oman, With EUCREAS® 50/1000 mg Tablets Manufactured by Novartis Pharma GmbH, Germany, in Normal, Healthy, Adult, Male Human Subjects Under Fed Conditions.
Brief Title: The Study Intends to Show Bioequivalence of the Test Product and the Reference Reference Product in a Crossover Design Study Healthy Volunteers. Additionally, the Safety Profile of Test Product Compared to Reference Product Will be Evaluated.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AET Laboratories Private Limited (Industry)
Responsible Party: Sponsor
Organization: Alfred E. Tiefenbacher (GmbH & Co. KG) (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 14-VIN-410
Record Dates: First submitted 2022-03-25; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: To Determine Bioequivalence Under Fed Conditions
MeSH Terms: interventions — Metformin; Vildagliptin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin and Vildagliptin 1000/50 mg Tablet (Experimental): 1 tablet of Metformin and Vildagliptin 1000/50 mg as single-dose administration
  Interventions: Drug: Metformin and Vildagliptin 1000/50 mg
- EUCREAS® 50/1000 mg Tablet (Active Comparator): 1 tablet of EUCREAS® 50/1000 mg (each film-coated tablet contains Vildagliptin 50 mg and Metformin hydrochloride 1000 mg) as single-dose administration
  Interventions: Drug: Metformin and Vildagliptin 1000/50 mg

INTERVENTIONS:
Drug: Metformin and Vildagliptin 1000/50 mg — 50 mg Vildagliptin + 1000 mg Metformin as single-dose per study period

SUMMARY:
To evaluate and compare the relative bioavailability and therefore the bioequivalence of fixed dose combination of Metformin and Vildagliptin Tablets 1000/50 mg manufactured by Oman Pharmaceuticals Products Co. LLC, Sultanate of Oman, with EUCREAS® 50/1000 mg tablets manufactured by Novartis Pharma GmbH, Germany, in Normal, Healthy, Adult, Male Human Subjects under Fed Conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged between 18 and 45 years (both inclusive).
2. Subjects' weight within the normal range according to normal values for the Body Mass Index (18.50 to 30.00 kg/m2) with minimum of 50 kg weight.
3. Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations within clinically acceptable normal range.
4. Subjects having clinically acceptable 12-lead electrocardiogram (ECG).
5. Subjects having clinically acceptable chest X-Ray (PA view).
6. Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine and morphine).
7. Subjects having negative alcohol breath test.
8. Subjects willing to adhere to the protocol requirements and to provide written informed consent.
9. No history or presence of smoking.
10. No history or presence of alcoholism and drug of abuse.

Exclusion Criteria:

1. Hypersensitivity to Vildagliptin or Metformin or related class of drugs.
2. History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
3. Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 1 month of the study starting.
4. History or presence of asthma, urticaria or other significant allergic reactions.
5. History or presence of significant gastric and/or duodenal ulceration.
6. History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
7. History or presence of cancer or basal or squamous cell carcinoma.
8. Difficulty with donating blood.
9. Difficulty in swallowing solids like tablets or capsules.
10. Use of any prescribed medication during the last one month or OTC medication during last two weeks prior to Dosing in Period 01.
11. Major illness during 3 months before screening.
12. Donation of blood in the past 3 months before screening.
13. Participation in drug research study within past 3 months.
14. Consumption of grapefruit juice within 72.00 hours prior to dosing in Period 01 and xanthine-containing products, tobacco containing products or alcohol within 48.00 hours prior to dosing in Period 01.
15. Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
16. History or presence of significant easy bruising or bleeding.
17. History or presence of significant recent trauma.
18. Subjects who have been on an abnormal diet (for whatever reason) during the four weeks preceding the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Cmax of Vildagliptin and Metformin for the test and reference products | up to 24 hours
  The maximum concentration in plasma among observed concentrations at pre-specified time points
AUC0-t of Vildagliptin and Metformin for the test and the reference products | up to 24 hours
  The area under the plasma concentration versus time curve from time 0 to the last measured concentration

SECONDARY OUTCOMES:
AUC0-∞ of Vildagliptin and Metformin for the test and the reference products | up to 24 hours
  The area under the plasma concentration versus time curve from time 0 to to infinite time
Tmax of Vildagliptin and Metformin for the test and the reference products | up to 24 hours
  The time to maximum measured plasma concentration
T1/2 of Vildagliptin and Metfomin for the test and the reference products | up to 24 hours
  Plasma elimination half-life
Kel of Vildagliptin and Metformin for the test and the reference products | up to 24 hours
  Elimination rate constant
Number of treatment-related adverse events (AE) for the test and the reference products as assessed by guidance predefined in the protocol | through study completion, an average of 1 month
  An AE is defined as any untoward medical occurrence in a subject administered the test or the reference product and which does not necessarily have a causal relationship with the treatment.